CLINICAL TRIAL: NCT05238415
Title: ASAP - Assisted Immediate Augmented Post-/Long-COVID Plan
Brief Title: ASAP - Assisted Immediate Augmented Post-/Long-COVID Plan for Patients Infected With COVID-19
Acronym: ASAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Sonia Lippke (Other)
Collaborators: Dr. Becker Hospital Group (Other); Dr. Becker Kiliani Clinic (Unknown); Dr. Becker Clinic Möhnesee (Unknown); Johannesbad Reha Clinics Bad Füssing (Unknown); Reha-Centre Bad Kötzting (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Dr. Sonia Lippke, Professor of Health Psychology and Behavioral Medicine, Jacobs University Bremen gGmbH
Organization: Jacobs University Bremen gGmbH (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: ASAP
Record Dates: First submitted 2022-02-10; First posted 2022-02-14 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Long-COVID; Post-COVID; Psychosomatic Disorder; Psychological Distress; Psychological Disease; Psychological Disorder; Psychological Impairment; Psychological Adjustment; Physiological Disease; Physiological Disorder; Physiological Impairment; Physiological Adjustment; Healthy Lifestyle
Keywords: Post-COVID; Long-COVID; treatment plan; eHealth; digital intervention; medical rehabilitation; psychosomatic rehabilitation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Psychophysiologic Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: This study has three study arms. Specifically, patients will be randomly assigned to an intervention group or an active control group. Furthermore, a comparison group will be recruited. Whereas the CompG will not receive any treatment, the IG and the ACG will have contacts with a personal pilot who will help the patients to navigate through the study as well as through treatment options and help them seek help for further needs. Aditionally, the intervention group will receive a so called 3-day assessment in a clinic and in which patients will be assessed by a multiprofessional team of health care professionals regarding their post-/long-COVID symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group receiving no Post-/Long-COVID assessment (No Intervention): Questionnaires at timepoints t1 (screening), t2 (one week later), t3 (before the intervention), t4 (after the intervention), t5 (6 weeks after intervention), t6 (6 months after the intervention)
  Patients from Bavaria Germany: Contact to personal pilots and digital health interventions.
- Intervention group receiving a Post-/Long-COVID assessment (Experimental): Questionnaires at timepoints t1 (screening), t2 (one week later), t3 (before the intervention), t4 (after the intervention), t5 (6 weeks after intervention), t6 (6 months after the intervention)
  Patients from Bavaria Germany: Assessment in clinics for post-/long-COVID, contact to personal pilots and digital health interventions.
  Interventions: Diagnostic Test: Psychological and Physiological Assessments
- Comparison group receiving no Post-/Long-COVID assessment (No Intervention): Questionnaires at timepoints t1 (screening), t2 (comparable to t2 in the other groups), t3 (comparable with t4 in the other groups), t3 (comparable to t5 in the other groups)
  Patients from Germany: No intervention at all

INTERVENTIONS:
Diagnostic Test: Psychological and Physiological Assessments — About N = 60 patients admitted to the study receive a 3-day assessment (a further examination) at the Kiliani-Klinik Bad Windsheim which considers physical and psychological parameters relevant for the diagnosis of a Post-/ Long-COVID Syndrom.
  Arms: Intervention group receiving a Post-/Long-COVID assessment

SUMMARY:
Post-/long-COVID occurs in patients with severe, moderate, and even mild courses. The symptomatology is multi-layered and complex. Patients with mild and moderate courses and especially younger patients are not optimally integrated into one of the existing care structures of COVID outpatient clinics and regular primary care. The diagnosis of post-/long-COVID and a consequent targeted treatment are currently partly not ensured. The variability of symptoms and the resulting complexity of diagnosis and treatment also pose a challenge in rural areas.

The aim of the project is an evaluation of a program for low-threshold needs identification and treatment planning for a hybrid (personal supporting counselors and digital trainings) post-/long-COVID care.

The contents of the present project include an innovative basis outside the existing standard care for the identification of affected persons. This will be done by means of a low-threshold online screening, which can also be carried out by the affected persons themselves. Furthermore, an intensive interdisciplinary assessment linked to medical rehabilitation resulting in a comprehensive, interdisciplinary, and cross-sectoral treatment plan is a core component of the current project. Finally, the implementation of digital trainings which are accompanied by a personal supporting counselor and augmented by continuously available trainings in the form of digital modules aim to provide general recommendation for the future support of post/long-COVID care.

The current research project aims to evaluate the feasibility and the practicability of a comprehensive, interdisciplinary, and cross-sectoral treatment program consisting of a low-threshold online screening and holistic assessment for PACS. Furthermore, it aims to evaluate digital interventions and the use of so-called personal guides that may help to facilitate the recovery of PACS.

DETAILED DESCRIPTION:
The goal is the long-term and sustainable holistic treatment and support of patients with post-/long-COVID to prevent long-term illness and chronification. Following the earliest possible, low-threshold identification of post-/long-COVID sufferers, an intensive multidisciplinary assessment is conducted, resulting in holistic treatment planning based on the results of the assessment. This consists of recommendations for a coordinated, interdisciplinary therapy plan. At the same time, digital therapy offers are recommended and made available to patients. Patients are accompanied by a supporting counselor (personal pilot) who guides them through the entire care process. This closes the gap between acute care of COVID-19 and outpatient therapy or rehabilitation of post-/long-COVID.

To identify patients with post-/long-COVID symptoms, a low-threshold scientifically based online-screening that confirms the presence of post-/long-COVID syndrome and an three day inpatient assessment that determines the need for further treatment will be developed, validated and prepared for standard care. Long-term goals are the dissemination of the validated instruments to diagnose post-long-COVID and treatment approaches (interdisciplinary, individualized treatment plan) through communication to key stakeholders such as medical associations, health insurance companies, service providers in the outpatient and inpatient sector, as well as professional societies and care institutions. This is intended to improve patient care and make care delivery of treatments for post-/long-COVID patients more efficient beyond the project duration.

Standard care currently diagnoses post-/long-COVID and provides recommendations for treatment through primary care practices and specialized post-COVID outpatient clinics. Both access routes inadequately reach those affected especially in rural areas. Long-/post-COVID outpatient clinics are primarily located in metropolitan areas and are therefore mainly available to the population in large cities. In particular, young affected individuals who have had little to no prior outpatient care due to a very mild course do not have primary care and often do not have the knowledge of the specific post-/long-COVID symptomatology and potentially seek insufficient and delayed medical support. This may result in aggravation and possibly chronification of symptoms and consequent long-term disability/ incapacity with limited participation. This in turn can have a negative impact on the continuation or resumption of work and lead to economic burdens for the whole society.

The contents of the present project include, as an innovative basis outside the existing standard care, the low-threshold identification of affected persons, an intensive interdisciplinary assessment resulting in a comprehensive, interdisciplinary and cross-sectoral treatment plan, the implementation of which is controlled and accompanied by a personal supporting counselor and augmented by continuously available training in the form of digital offers.

The following research questions and hypotheses will be investigated with this project and subsequently communicated to the various stakeholders and the general public:

1. What screening tool can reliably identify patients suffering from post/long-COVID syndrome? Hypothesis: With a simplified screening, the presence of post/long-COVID can be identified in a low-threshold manner.
2. Which assessments can be used to reliably determine the need for therapy or rehabilitation and the leading rehabilitation indication? Hypothesis: With a comprehensive assessment, the need for rehabilitation and the leading rehabilitation indication can be determined validly and reliably.
3. What must digital therapy offerings look like to benefit patients with post/long-COVID syndrome? Hypothesis: Digital therapy offerings with an individualizable focus achieve the best success in the treatment of post/long-COVID.
4. What information must the supporting counselor have to ensure management of interdisciplinary treatment? Hypothesis: As a point of contact for all stakeholders, a supporting counselor will have interdisciplinary and intersectoral treatment planning available to ensure sustained management of interdisciplinary treatment.
5. How should an interdisciplinary treatment pathway look like in the long term? Hypothesis: An interdisciplinary treatment pathway must guide the patient, with the support of the supporting counselor, in such a way that he or she experiences the appropriate diagnosis and treatment for him or herself and actively participates in recovery so that he or she recovers quickly and sustainably from his or her post/long-COVID disease, increases his or her functional capacity, reduces incapacity to work, and regains participation.

The project aims to optimize care for post-/long-COVID patients and empower them to participate socially. Affected individuals are supported on their way to the appropriate therapeutic and rehabilitative care by expert staff, the supporting counselors (personal pilots), and receive interdisciplinary multi-professional treatment focused on individual complaints. Affected individuals are accompanied and supported through digital interventions. The low-threshold access via an online-screening leads to the elimination of information loss and inhibitions. Various digital services, such as DiGAs, video consultations, as well as aftercare services are increasingly used. This is of particular benefit to patients who have tight schedules and/or live in rural regions with a low density of doctors/therapists.

ELIGIBILITY:
Inclusion Criteria:

* All people who are resident in Bavaria can participate in the intervention and control group. In the comparison group all people who live and work in Germany can take part
* working age
* ability to participate in surveys (e.g., sufficient German language skills)
* willingness to participate in outpatient or (partially) inpatient therapy
* ability to undergo rehabilitation if necessary, and a telephone and Internet connection
* suspicion of post-/long-COVID

Exclusion Criteria:

* Contraindications regarding physical exercise,
* not being of age,
* illiteracy
* massively limited cognitive abilities (linguistic components of the digital offerings must be able to be used and questionnaires completed or interviews participated in)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Post-/ Long-COVID symptoms at 3 months | Baseline to 3 months
  The symptom change with regard to Post-/Long-COVID will be evaluated by at least three follow-up measures, using a questionnaire adapted from the COVID-19 Rehabilitation Needs Questionnaire-Health Problems caused by SARS-CoV-2 (Lemhöfer, C., et al. (2021)), with 14 items. Possible scores range from 1 (no problem) to 5 (extreme problem). Change = (Score at measurement points (e.g.,3 months) - Score at baseline)
Subjective prognosis of return to work | 2 weeks, 8 weeks
  Return to work will be evaluated by at least one follow-up measure, e.g., T2 (2 weeks from baseline), T4 (8 weeks from baseline). The questionnaire is adapted to the context of COVID-19 from the SPE scale (Mittag, O., & Raspe, H. (2003)), with 4 items.

SECONDARY OUTCOMES:
Activity and social participation | 2 weeks, 8 weeks
  Social participation will be evaluated by at least one follow-up measure, e.g., T2 (2 weeks from baseline), T4 (8 weeks from baseline), using a questionnaire adapted from the COVID-19 Rehabilitation Needs Questionnaire-Activity and participation (Lemhöfer, C., et al. (2021)), with 12 items. Possible scores range from 1 (Never) to 5 (Often/always).
Health behaviors of daily living | 2 weeks, 8 weeks
  Health behaviors of daily living including physical activity and nutrition consumption behavior, and sedentary behavior will be evaluated by at least one follow-up measure, e.g., T2 (2 weeks from baseline), T4 (8 weeks from baseline). The physical activity and nutrition consumption questionnaire is adapted from the Physical Activity and Fruit and Vegetable Consumption Questionnaire (Lippke, S., et al. (2009)), with 2 items. The sedentary behavior questionnaire is adapted from the International Physical Activity Questionnaire (Craig, C. L.,et al. (2003)), with 2 Items.
Mental health | 2 weeks, 8 weeks
  Mental health including loneliness, psychological distress, stress, depression and anxiety will be evaluated by at least one follow-up measure, e.g., T2 (2 weeks from baseline), T4 (8 weeks from baseline). The loneliness questionnaire is adapted from the UCLA loneliness scale (Russell, D. (1996)), with 2 items. The psychological distress will be assessed by Peri-traumatic Distress Scale (Qiu, J. et al. (2020)), with 24 items. The stress questionnaire is adapted from the PSS-4 (Cohen, S. (1988)), with 4 items. The depression and anxiety questionnaire is adapted from the PHQ-4 (Löwe, B.,et al. (2010)), with 4 items.
Life satisfaction | 2 weeks, 8 weeks
  Life satisfaction will be evaluated by at least one follow-up measure, e.g., T2 (2 weeks from baseline), T4 (8 weeks from baseline), using a questionnaire adapted from the General Satisfaction with Life Questionnaire (Beierlein, C., et al. (2015)), with 4 items. Possible scores range from 1 (totally unsatisfied) to 4 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, Prof. Dr., Principal Investigator — Jacobs University Bremen
Locations (1):
- Dr. Becker Klinikgruppe, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be published. Other researchers are welcome to get in contact with the PI to get access to anonymous data.

REFERENCES:
- [Background] Akhmerov A, Marban E. COVID-19 and the Heart. Circ Res. 2020 May 8;126(10):1443-1455. doi: 10.1161/CIRCRESAHA.120.317055. Epub 2020 Apr 7. PMID 32252591
- [Background] Cai X, Hu X, Ekumi IO, Wang J, An Y, Li Z, Yuan B. Psychological Distress and Its Correlates Among COVID-19 Survivors During Early Convalescence Across Age Groups. Am J Geriatr Psychiatry. 2020 Oct;28(10):1030-1039. doi: 10.1016/j.jagp.2020.07.003. Epub 2020 Jul 10. PMID 32753338
- [Background] - Dahmen A, Gao L, Keller FM, Becker P & Lippke S. Psychosomatische Nachsorge: Curriculum Hannover online vs. Curriculum Hannover und vs. Care as Usual. Vortrag im Rahmen des DRV-Kolloquiums 2021.
- [Background] - Dahmen A & Becker P. Abschlussbericht des Umsetzungsprojektes Curriculum Hannover-Online - Studien zur Wirksamkeit und Äquivalenz einer internetbasierten Virtual-Classroom-Intervention zur psychosomatischen Nachsorge nach dem Curriculum Hannover, o.a.
- [Background] - DIMDI. ICF - Internationale Klassifikation der Funktionsfähigkeit, Behinderung und Gesundheit. WHO, Genf, 2005.
- [Background] - Gutenbrunner C et al., Rehabilitation bei und nach SARS-CoV-2 Infektionen. das Krankenhaus 112 (2021): 02.
- [Background] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Background] - Kassenärztliche Bundesvereinigung (KBV). Versichertenbefragung der Kassenärztlichen Bundesvereinigung 2021. FGW Forschungsgruppe Wahlen Telefonfeld GmbH, Mannheim, 2021.
- [Background] Keller FM, Dahmen A, Derksen C, Kotting L, Lippke S. Psychosomatic Rehabilitation Patients and the General Population During COVID-19: Online Cross-sectional and Longitudinal Study of Digital Trainings and Rehabilitation Effects. JMIR Ment Health. 2021 Aug 26;8(8):e30610. doi: 10.2196/30610. PMID 34270444
- [Background] - Klapsa, K. Die Angst, dass Long-COVID-Patienten das Gesundheitssystem überfordern. https://www.welt.de/politik/deutschland/article230250123/Rehakliniken-Erleben-massive-Zunahme-von-Long-Covid-Patienten.html, 16.04.2021 (Zugriff am: 14.09.2021)
- [Background] - Kluge et al., S3-Leitlinie - Empfehlungen zur stationären Therapie von Patienten mit COVID-19. AWMF-Register Nr. 113/001, 2021.
- [Background] - Koczulla AR et al. S1-Leitlinie Post-COVID/Long-COVID, AWMF-Register Nr. 020/027, 2021.
- [Background] Mazza C, Ricci E, Biondi S, Colasanti M, Ferracuti S, Napoli C, Roma P. A Nationwide Survey of Psychological Distress among Italian People during the COVID-19 Pandemic: Immediate Psychological Responses and Associated Factors. Int J Environ Res Public Health. 2020 May 2;17(9):3165. doi: 10.3390/ijerph17093165. PMID 32370116
- [Background] Nalbandian A, Sehgal K, Gupta A, Madhavan MV, McGroder C, Stevens JS, Cook JR, Nordvig AS, Shalev D, Sehrawat TS, Ahluwalia N, Bikdeli B, Dietz D, Der-Nigoghossian C, Liyanage-Don N, Rosner GF, Bernstein EJ, Mohan S, Beckley AA, Seres DS, Choueiri TK, Uriel N, Ausiello JC, Accili D, Freedberg DE, Baldwin M, Schwartz A, Brodie D, Garcia CK, Elkind MSV, Connors JM, Bilezikian JP, Landry DW, Wan EY. Post-acute COVID-19 syndrome. Nat Med. 2021 Apr;27(4):601-615. doi: 10.1038/s41591-021-01283-z. Epub 2021 Mar 22. PMID 33753937
- [Background] - National Institute of Health, NIH Plans Research on "Long COVID". https://covid19.nih.gov/news-and-stories/research-on-long-covid, 2021.
- [Background] Paterson RW, Brown RL, Benjamin L, Nortley R, Wiethoff S, Bharucha T, Jayaseelan DL, Kumar G, Raftopoulos RE, Zambreanu L, Vivekanandam V, Khoo A, Geraldes R, Chinthapalli K, Boyd E, Tuzlali H, Price G, Christofi G, Morrow J, McNamara P, McLoughlin B, Lim ST, Mehta PR, Levee V, Keddie S, Yong W, Trip SA, Foulkes AJM, Hotton G, Miller TD, Everitt AD, Carswell C, Davies NWS, Yoong M, Attwell D, Sreedharan J, Silber E, Schott JM, Chandratheva A, Perry RJ, Simister R, Checkley A, Longley N, Farmer SF, Carletti F, Houlihan C, Thom M, Lunn MP, Spillane J, Howard R, Vincent A, Werring DJ, Hoskote C, Jager HR, Manji H, Zandi MS. The emerging spectrum of COVID-19 neurology: clinical, radiological and laboratory findings. Brain. 2020 Oct 1;143(10):3104-3120. doi: 10.1093/brain/awaa240. PMID 32637987
- [Background] - Schlitt A, Schultz K, Platz T. AWMF-Leitlinie: Rehabilitation nach einer COVID-19-Erkrankung. Dtsch Ärztebl 2021; 118: A774.
- [Background] - Schmädeke S et al. Abschlussbericht des Umsetzungsprojekts Rehabilitationsnachsorge für depressive Patientinnen und Patienten mit einer Smartphone-App (DE-RENA) - Akzeptanz, Wirksamkeit und Empfehlungen, o.a.
- [Background] Seecheran R, Narayansingh R, Giddings S, Rampaul M, Furlonge K, Abdool K, Bhagwandass N, Seecheran NA. Atrial Arrhythmias in a Patient Presenting With Coronavirus Disease-2019 (COVID-19) Infection. J Investig Med High Impact Case Rep. 2020 Jan-Dec;8:2324709620925571. doi: 10.1177/2324709620925571. PMID 32370558
- [Background] Venkatesan P. NICE guideline on long COVID. Lancet Respir Med. 2021 Feb;9(2):129. doi: 10.1016/S2213-2600(21)00031-X. Epub 2021 Jan 13. No abstract available. PMID 33453162
- [Background] - WIdO, Ein Jahr Covid-19-bedingte Fehlzeiten am Arbeitsplatz: Jeder zwölfte betroffene Beschäftigte musste stationär behandelt werden, Pressemitteilung, 2021.
- [Background] - Wolf, S. and Erdös, J. for the Belgian Health Care Knowledge Centre (KCE). Epidemiology of long COVID: a preliminary report. Deutsche Kurzfassung zum gleichnamigen KCE-Bericht. AIHTA Projektbericht Nr. 135a; 2021. Wien: Austrian Institute for Health Technology Assessment GmbH.
- [Derived] Derksen C, Rinn R, Gao L, Dahmen A, Cordes C, Kolb C, Becker P, Lippke S. Longitudinal Evaluation of an Integrated Post-COVID-19/Long COVID Management Program Consisting of Digital Interventions and Personal Support: Randomized Controlled Trial. J Med Internet Res. 2023 Oct 4;25:e49342. doi: 10.2196/49342. PMID 37792437
- [Derived] Dahmen A, Keller FM, Derksen C, Rinn R, Becker P, Lippke S. Screening and assessment for post-acute COVID-19 syndrome (PACS), guidance by personal pilots and support with individual digital trainings within intersectoral care: a study protocol of a randomized controlled trial. BMC Infect Dis. 2022 Aug 15;22(1):693. doi: 10.1186/s12879-022-07584-z. PMID 35971066
- See also: 10.08.2021 — http://www.aerztezeitung.de/Nachrichten/Holetschek-Post-COVID-Erkrankungen-haben-Potenzial-zur-Volkskrankheit-421867.html
- See also: 09.08.2021 — http://www.aerztezeitung.de/Nachrichten/Neue-Corona-Studien-Remdesivir-Lockdown-Folgen-Masken-et-al-410212.html
- See also: 12.08.2021 — http://www.rki.de/DE/Content/InfAZ/N/Neuartiges_Coronavirus/Teststrategie/Nat-Teststrat.html
- See also: 12.08.2021 — http://www.aerzteblatt.de/nachrichten/125092/Neue-neurologisch-psychiatrische-Post-COVID-Ambulanz-in-Muenchen